CLINICAL TRIAL: NCT01833767
Title: Phase 2 Trial of T-cell Based Low-dose Cyclophosphamide and Outpatient Intravenous Interleukin-2 in Metastatic Melanoma
Brief Title: Low-dose Cyclophosphamide and Outpatient IV Interleukin-2 in Metastatic Melanoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Principal Investigator, Jordan Waypa, Research Director, Western Regional Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-12
Record Dates: First submitted 2013-04-14; First posted 2013-04-17 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cyclophosphamide and Interleukin-2 (Experimental): Cytoxan IV on day 1, IL2 IV on days 1-5
  Interventions: Drug: Cyclophosphamide and Interleukin 2

INTERVENTIONS:
Drug: Cyclophosphamide and Interleukin 2 — Cytoxan IV day 1, IL2 IV days 1-5
  Other Names: Cytoxan; IL2

SUMMARY:
The purpose of this study is to determine response rates by administering low dose cyclophosphamide on day 1, followed by 5 days of outpatient IL2.

DETAILED DESCRIPTION:
To determine the response rate, median duration of response and median survival of patients treated with this low-dose cyclophosphamide + moderate dose bolus Interleukin-2 schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologic diagnosis of metastatic melanoma. Patients may have received prior systemic therapy or may be previously untreated.
2. Patients must have measurable disease on physical exam or radiologic studies.
3. ECOG performance status of 0 or 1 and estimated survival of at least 3 months.
4. White blood count of > 3500/mm3, platelet count > 100,000/mm3, hemoglobin > 9.0 gm/dl; bilirubin, ALT, AST < 3 x upper limit of normal; serum creatinine < 2.0 mg/dl.
5. Patients must undergo a low-level cardiac stress test as a screen for possible atherosclerotic heart disease. Patients with a positive stress test would be excluded from this trial.
6. Patients with elevated temperatures > 100.5 F must have sources of occult infection excluded.
7. Patients must be felt to have recovered from effects of prior therapy, such as > 2 weeks after prior chemotherapy.
8. Women of childbearing potential must have a negative pregnancy test and adequate precautions to prevent pregnancy during treatment must be taken.
9. Patient consent must be obtained prior to entrance onto study.

Exclusion Criteria:

* 1. Medical illness requiring corticosteroids or other immunosuppressive agents (such as cyclosporin or methotrexate.

  2. Autoimmune disease such as inflammatory arthritis which could be exacerbated by immune-based therapy.

  3. Prior history of psychiatric disorder which could be exacerbated by interleukin-2.

  4. Lactation or pregnancy.

  5. Evidence of significant cardiovascular disease including history of recent (< 6 months prior) myocardial infarction, congestive heart failure, primary cardiac arrhythmias (not due to electrolyte disorder or drug toxicity, for example) beyond occasional PVC's, angina, positive low-level stress test, or cerebrovascular accident.

  6. Current untreated brain metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Response Rate | One year

SECONDARY OUTCOMES:
Median Survival | One year

CONTACTS AND LOCATIONS:
Overall Officials: Walter Quan, MD, Principal Investigator — Western Regional Medical Center
Locations (1):
- Western Regional Medical Center Inc, Goodyear, Arizona, United States